CLINICAL TRIAL: NCT01098097
Title: Post Marketing Observational/Non-Interventional Study Of Retreatment Of Chronic Hepatitis C With Peginterferon Alpha And Ribavirin
Brief Title: Post Marketing Observational Study of Retreatment of Chronic Hepatitis C With Peginterferon Alpha and Ribavirin (Study P06011)
Acronym: POMOSCH
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P06011
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Results first posted 2012-11-20 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peginterferon alpha and ribavirin: Peginterferon alpha and ribavirin will be administered at the discretion of the treating physician, in accordance per label according to local guidelines for all participating countries.
  Interventions: Biological: Peginterferon alpha; Drug: Ribavirin

INTERVENTIONS:
Biological: Peginterferon alpha — Peginterferon alpha given in combination with ribavirin according to local labeling guidelines
  Other Names: PegIntron; SCH 054031; MK-4031
Drug: Ribavirin — Ribavirin given in combination with peginterferon alpha according to local labeling guidelines
  Other Names: Rebetol; SCH 018908; MK-8908

SUMMARY:
To study retreatment in patients who failed prior treatment with interferon alpha (pegylated or non-pegylated) with or without ribavirin in a real-life setting in an observational/noninterventional study.

DETAILED DESCRIPTION:
This is an observational/non interventional study to collect data on the patient characteristics of those seeking retreatment as well as safety and efficacy information during the first 12 weeks of retreatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C of any genotype;
* Prior treatment with interferon alpha (pegylated or non-pegylated) with or without ribavirin did not result in a sustained virological response;
* Inclusion criteria listed on the approved label in each country;
* Willingness of the patient to participate and sign the Informed Consent Form.

Exclusion Criteria:

* Patient exclusion from this observational/non-interventional study will be determined by the treating physician and will be based on the local label in each country.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who failed prior treatment with interferon alpha (pegylated or non-pegylated) with or without ribavirin
Sampling Method: Non-Probability Sample
Enrollment: 963 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled: 9 February 2009; last participant completed: 17 October 2011. The study was conducted in 117 centers in 12 countries.
Groups:
- Peginterferon Alpha and Ribavirin: Peginterferon alpha and ribavirin was administered at the discretion of the treating physician, in accordance per label according to local guidelines for all participating countries.
Period: Overall Study
Arm/Group | Peginterferon Alpha and Ribavirin
Started | 963
Completed | 881 (Participants completing the study received at least 12 weeks of treatment)
Not Completed | 82
Not completed — Adverse Event | 17
Not completed — Lost to Follow-up | 18
Not completed — Status unknown | 16
Not completed — No reason reported | 31

BASELINE CHARACTERISTICS:
Arm/Group | Peginterferon Alpha and Ribavirin
Number analyzed (Participants) | 963
Age, Continuous [Median (Full Range); unit: years] | 50 [18 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 420
  Male | 543
Previous non-response type [Number; unit: participants] — Participants in the study previously failed to respond with a sustained virologic response to treatment with interferon alpha with or without ribavirin. The type of previous non-response was categorized at study baseline.
  participants
    Null responder | 346
    Virologic breakthrough | 67
    Relapse | 544
    Previous non-response type not known | 6

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Serious Adverse Events (SAEs) and/or Clinically Significant Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product which did not necessarily have a causal relationship to the treatment. All AEs reported in the study were judged by the investigator to be clinically significant. An SAE was any adverse drug experience that resulted in death, was life-threatening, caused or prolonged hospitalization, caused persistent or significant disability or incapacity, caused a congenital anomaly or birth defect, or may have required medical or surgical intervention to prevent one of these outcomes.
Time Frame: Up to 12 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alpha and Ribavirin
Number analyzed (Participants) | 963
percentage of participants
  Clinically significant adverse event | 33.6
  Serious adverse event | 1.9

2. Primary Outcome: Incidence of Thrombocytopenia
Description: Thrombocytopenia is a low blood platelet count
Time Frame: Up to 12 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alpha and Ribavirin
Number analyzed (Participants) | 963
percentage of participants | 3.8

3. Primary Outcome: Incidence of Treatment Discontinuations Due to Adverse Events
Description: All treatment discontinuations due to an AE were reported. See Outcome Measure 1 for definition of AEs.
Time Frame: Up to 12 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alpha and Ribavirin
Number analyzed (Participants) | 963
percentage of participants
  Treatment stopped - any AE | 2.6
  Dose reduced, then treatment stopped - any AE | 0.1

4. Primary Outcome: Incidence of Particular Adverse Events Resulting in Treatment Discontinuation
Description: All treatment discontinuations due to particular AEs were reported. These discontinuations included treatment stopped (TS) and dose reduced followed by treatment stopped (DR/TS).
  The particular AE evaluated were anemia (low red blood cells), leucopenia (low white blood cells), neutropenia (low blood neutrophils), thrombocytopenia (low blood platelets), esophageal varices (dilated veins in lower esophagus), splenomegaly (enlarged spleen), portal hypertensive gastropathy (changes in stomach mucosa), and hepatomegaly (enlarged liver)
Time Frame: Up to 12 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alpha and Ribavirin
Number analyzed (Participants) | 963
percentage of participants
  TS - Anemia | 0.6
  TS - Leucopenia | 0.2
  TS - Neutropenia | 0.2
  TS - Thrombocytopenia | 0.1
  TS - Esophageal varices | 0.0
  TS - Splenomegaly | 0.0
  TS -Portal hypertensive gastropathy | 0.0
  TS - Hepatomegaly | 0.0
  DR/TS - Anemia | 0.1
  DR/TS - Leucopenia | 0.0
  DR/TS - Neutropenia | 0.0
  DR/TS - Thrombocytopenia | 0.0
  DR/TS - Esophageal varices | 0.0
  DR/TS - Splenomegaly | 0.0
  DR/TS - Portal hypertensive gastropathy | 0.0
  DR/TS - Hepatomegaly | 0.0

5. Primary Outcome: Incidence of Dose Modifications Due to Adverse Events
Description: All dose modifications due to an AE were reported. See Outcome Measure 1 for definition of AEs.
Time Frame: Up to 12 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alpha and Ribavirin
Number analyzed (Participants) | 963
percentage of participants
  Dose Reduced | 9.7
  Dose Reduced, then Treatment Stopped | 0.1
  Dose Reduced, Treatment Suspended and Restarted | 0.3

6. Secondary Outcome: Proportion of Participants Who Achieve Undetectable Hepatitis C Virus Ribonucleic Acid (HCV-RNA)
Description: Participant's blood was tested for HCV-RNA by quantitative polymerase chain reaction. The limit of detection for the assay was 50 IU/mL.
Time Frame: Week 12
Population: The population analyzed was 920 participants who received at least 1 dose of study drug and had data collected at the Week 12 visit
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peginterferon Alpha and Ribavirin
Number analyzed (Participants) | 920
percentage of participants | 42.4 [39.1 to 45.9]

ADVERSE EVENTS:
Arm/Group | Peginterferon Alpha and Ribavirin
Serious Adverse Events (participants affected / at risk) | 18/963
Other Adverse Events (participants affected / at risk) | 211/963
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon Alpha and Ribavirin (N=963)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Leucopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Acute tonsillitis (Infections and infestations) | 1 (1)
Campylobacter infection (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon Alpha and Ribavirin (N=963)
Anaemia (Blood and lymphatic system disorders) | 104 (106)
Leucopenia (Blood and lymphatic system disorders) | 52 (55)
Neutropenia (Blood and lymphatic system disorders) | 55 (59)
Fatigue (General disorders) | 49 (49)
Pyrexia (General disorders) | 54 (59)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts. Investigator agrees to meet with sponsor's representatives prior to submission for publication to discuss and resolve any disagreements.